CLINICAL TRIAL: NCT03165474
Title: Intervention INC: Interactive Nutrition Comics for Urban Minority Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter College of City University of New York (Other)
Collaborators: Children's Aid (Unknown); Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Device Feasibility
Other Study IDs: HunterCCUNY
Record Dates: First submitted 2017-05-15; First posted 2017-05-24 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Obesity, Childhood
Keywords: childhood obesity; mhealth; digital health; nutrition; intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be randomized into intervention or control arm and will be provided with different orientations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Arm (Active Comparator): In the control group, children and parents will receive didactic health information and resources by email and/or text. The delivery mode of the health messages will be based on based on personal preference.
  Interventions: Other: Didactic health information
- Intervention Arm (Experimental): In the intervention group, children will have access to a web-based interactive nutrition comic and receive health messages from comic characters by email and/or text, while parents will receive weekly newsletters related to nutrition and health by email and/or text.
  Interventions: Other: Web-based comic and newsletters

INTERVENTIONS:
Other: Web-based comic and newsletters — Web-based comic and health messages (child component) and health newsletters (parent component)
  Arms: Intervention Arm
Other: Didactic health information — Didactic health information and resources by email and/or text
  Arms: Control Arm

SUMMARY:
The primary purpose of this study is to assess the feasibility and participant acceptability of an interactive, internet/mobile-enabled dietary self management intervention. The secondary purpose of this study is to determine if the intervention improves knowledge, attitudes and food preferences associated with the targeted behaviors, to reduce childhood obesity risk from baseline to post-test.

DETAILED DESCRIPTION:
Based on inclusion/exclusion criteria, potential study participants (child and parent) will be identified by the Collaborating Site PI/primary contact and sent a recruitment letter signed by the Primary Investigator and a Collaborating Site PI/primary contact.

Children's Aid Society (CAS) and Weill Cornell Medical College (WCMC) will act as collaborating sites. WCMC PI is Dr. Allison Gorman, who will assist with identifying potential study participants from their government insured medical clinics. All recruitment protocols will be approved by the IRB at WCMC (pending Hunter IRB approval). Once the letter of approval has been received from WCMC, it will be forwarded to CUNY's HRPP. CAS primary contact is Alyson Abrami. Ms. Abrami and the CAS Milbank Medical Clinic will facilitate access to potential study participants. CAS is aware of the study protocols and the administration is in support of the study and its potential impact on their patient population.

Study staff will contact potential study participants by phone and ask additional screening questions to determine study eligibility. A baseline in-person study visit will be scheduled for eligible participants. We are aiming to recruit a total of 82 child/parent dyads (41 in the intervention and control group, respectively). In the intervention group, children will have access to a web-based interactive nutrition comic and receive health messages from comic characters by email and/or text, while parents will receive weekly newsletters related to nutrition and health by email and/or text. In the control group, children and parents will receive didactic health information and resources by email and/or text. The delivery mode of the health messages will be based on based on personal preference.

Aside from usage data of the online tool by each child/parent (e.g. average time spent per login using online tool, collected on an ongoing basis throughout 6-week intervention), data will be collected at four different times points in the study: baseline (T1), after 3 weeks or halfway through the intervention (T2-only children), after 6 weeks or at the end of the intervention (T3), and 3 months post-intervention (T4). T1 and T4 will be in-person study visits at either CUNY Hunter College or CAS Milbank. At baseline (T1), the child's height and weight will be measured to confirm meeting BMI eligibility criteria. After the child and parent completes consent/assent forms, they will be randomized to either the intervention group or control group. Both the child and parent will complete baseline survey measures (will take 20-30 minutes to complete) and attend a study orientation session (10-15 minutes). The baseline visit should take about 1 hour. At T2 (child-only) and T3 (child and parent), data collection (survey measures and open-ended questions) will be conducted either on the phone or by videochat in a private area, according to the participant preference, and will take approximately 30 minutes per person. At T4, the child's height and weight will be measured, and both the child and parent will complete survey measures (will take approximately 45 minutes to complete). Both the child and parent will be compensated for completing survey measures (see Participants-Compensation section for more details).

Open-ended questions collected at timepoint T3 (over the phone or videochat) will be audio recorded (only intervention arm participants). Even though participants will have signed consent to be audio recorded during data collection, the participant will be asked during the phone call or videochat session at T3 if the following open-ended questions could be audio recorded to be reviewed in more detail afterwards. Additionally, open-ended questions related to the experience and context of using the web-based nutrition comic will be asked of a subset of parents and children (intervention arm only) at timepoint T3 (over the phone or videochat). Their responses will also be audio recorded as this is qualitative data that will be transcribed and analyzed separately from survey data.

ELIGIBILITY:
Child Inclusion Criteria:

* Identify as Black, African-American, and/or Hispanic/Latino
* age 9-12 years old by start of the intervention
* English-speaking
* either received care at the WCMC clinic or CAS Milbank clinic within the last 2 years -
* has BMI percentile at or above 5% as indicated in their electronic health record (based on CDC sex-specific BMI-for-age- growth chart)
* has regular internet access via tablet, smartphone, and/or computer/laptop
* has regular phone access with texting ability
* has no allergies, food aversions, food disorders, or medications with side-effects that impact diet/eating that would prevent participation in the study
* has a parent/guardian willing to participate in the study

Parent inclusion criteria:

* Parent or guardian of child that meets inclusions/exclusion criteria
* English- or Spanish-speaking
* has regular internet access via tablet, smartphone, and/or computer/laptop
* has regular phone access with texting ability
* willing and able to give permission for their child to participate in the study

Exclusion Criteria:

* Participants involved in Aim 1 or Aim 2 of study previously exposed to components of intervention

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 178 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Usage - Child | Daily throughout study duration (~4.5 months)
  Usage analytics measured at the individual-level: min, max, average logins per day/week; min, max, average time spent on website per login; min, max, average link clicks per session (links to unique website areas)
Usability - Child | T2 (after 3 weeks or halfway through the intervention) and T3 (after 6 weeks or at the end of the intervention)
  Survey measure to assess usability, usefulness, ease of use, ease of learning, and satisfaction (taken from SUS, USE, and SUPR-Q survey)
Context of Use - Child | T3 (after 6 weeks or at the end of the intervention)
  Open-ended questions regarding experience and context using the web app, as well as acceptability and satisfaction

SECONDARY OUTCOMES:
Change in child knowledge & attitudes - Child | T1 (baseline), T2 (after 3 weeks or halfway through the intervention), T3 (after 6 weeks or at the end of the intervention),T4 (3 months post-intervention)
  Survey measuring change in child knowledge, self-efficacy, preferences, and outcome expectancies related to eating fruits/vegetables and consuming water
Change in child dietary intake - Child | T1 (baseline), T3 (after 6 weeks or at the end of the intervention),T4 (3 months post-intervention)
  Survey measuring change in child intake of specified fruits/vegetables, and water
Change in BMI percentile - Child | T1 (baseline) and T4 (3 months post-intervention)
  Change in BMI percentile calculated based on measured height and weight
Usage - Parent | Daily throughout study duration (~4.5 months)
  Usage analytics measured at the individual-level: min, max, average logins per day/week; min, max, average time spent on website per login; min, max, average link clicks per session (links to unique website areas)
Change in parent feeding practices - Parent | T1 (baseline), T3 (after 6 weeks or at the end of the intervention),T4 (3 months post-intervention)
  Survey measuring child involvement, parent encouragement, parent modeling, and parent instruction about fruits/vegetables and water intake
Change in physical home food environment | T1 (baseline), T3 (after 6 weeks or at the end of the intervention),T4 (3 months post-intervention)
  Survey measuring home availability and accessibility of fruits/vegetables and water

CONTACTS AND LOCATIONS:
Overall Officials: May May Leung, PhD, RDN, Principal Investigator — Hunter College of City University of New York
Locations (1):
- Hunter College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung MM, Mateo KF, Dublin M, Harrison L, Verdaguer S, Wyka K. Testing a Web-Based Interactive Comic Tool to Decrease Obesity Risk Among Racial and Ethnic Minority Preadolescents: Randomized Controlled Trial. JMIR Form Res. 2025 Jan 15;9:e58460. doi: 10.2196/58460. PMID 39813083
- [Derived] DeFrank G, Singh S, Mateo KF, Harrison L, Rosenthal A, Gorman A, Leung MM. Key recruitment and retention strategies for a pilot web-based intervention to decrease obesity risk among minority youth. Pilot Feasibility Stud. 2019 Sep 5;5:109. doi: 10.1186/s40814-019-0492-8. eCollection 2019. PMID 31516726
- [Derived] Leung MM, Mateo KF, Verdaguer S, Wyka K. Testing a Web-Based Interactive Comic Tool to Decrease Obesity Risk Among Minority Preadolescents: Protocol for a Pilot Randomized Control Trial. JMIR Res Protoc. 2018 Nov 9;7(11):e10682. doi: 10.2196/10682. PMID 30413399